CLINICAL TRIAL: NCT00634595
Title: A Randomized Phase II Clinical Trial of an Adenovirus-mediated Endostatin Gene (E10A) Combined With Cisplatin and Paclitaxel in Patients With Head and Neck Cancer
Brief Title: Trial of E10A in Head and Neck Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: Doublle Bioproduct Inc (Industry)
Responsible Party: Wenqi Jiang, Professor, Cancer center, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TG0717E10A
Record Dates: First submitted 2008-03-05; First posted 2008-03-13 (Estimated); Last update posted 2010-07-28 (Estimated); Status verified 2010-07

CONDITIONS: Head and Neck Squamous Carcinoma; Nasopharyngeal Carcinoma
Keywords: clinical trial; randomized; Endostatin; gene therapy; head and neck cancer; head and neck squamous carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma; Head and Neck Neoplasms | interventions — Cisplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): E10A combined with Cisplatin and Paclitaxel
  Interventions: Drug: E10A; Drug: Cisplatin; Drug: Paclitaxel
- B (Active Comparator): Cisplatin and Paclitaxel
  Interventions: Drug: Cisplatin; Drug: Paclitaxel

INTERVENTIONS:
Drug: E10A — E10A 1*10(12)VP, intratumoral injection, d1 d8, repeat every 3 weeks for 4 cycles
  Arms: A
Drug: Cisplatin — 25 mg/m2/d ivd d3 d4 d5, repeat every 3 weeks for 4 cycles.
Drug: Paclitaxel — 160 mg/m2 ivd d3, repeat every 3 weeks for 4 cycles.

SUMMARY:
Angiogenesis, the formation of new blood vessel from existing vessels, is essential for tumor growth and metastasis. Antiangiogenic therapies inhibit the growth of genetically stable endothelial cells, and most tumors should starve to death with little acquired resistance. Endostatin has been shown to block endothelial cell proliferation, survival, and migration. Antitumor activity of endostatin protein has been demonstrated in various murine and human tumors in animal model studies without any detectable toxicity. Endostatin gene therapy could directly express the highly bioactive protein in vivo by means of the mechanism of eukaryotic expression system as post-translational modification and folding, as well as overcoming the challenge of the long-term storage and the cumbersome daily administration of endostatin protein.

E10A is a replication-deficient recombinant adenovirus containing a wild-type human endostatin transgene constructed from serotype 5 adenovirus (Ad5). Preclinical studies demonstrated that intratumoral injection of E10A provided significant tumor growth inhibition and sustained elevation of endostatin in blood and tumor tissue in hepatocellular carcinoma, nasopharyngeal carcinoma, and tongue cancer animal models. A Phase I clinical trial of E10A we conducted showed that repetitive intratumoral injection of E10A resulted in a small and sustained elevation of endostatin in blood and had a mild antitumor activities with very limited toxicity. The major toxicity was transient and manageable fever. A randomized Phase III trial in nonsmall-cell lung cancer showed endostatin improved response rate and time to tumor progression in combination to chemotherapy. Therefore, we designed a randomized phase II trial to explore the safety and effectiveness of E10A combined with chemotherapy in the treatment of patients with head and neck cancer.

ELIGIBILITY:
Inclusion Criteria:

* histologically or cytologically confirmed recurrent or metastatic head and neck squamous carcinoma or nasopharyngeal carcinoma
* the tumor was amenable to direct injection and measurement ( > 2 cm)
* an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2
* a life expectancy over three months
* the absence of serious medical or psychiatric disorders
* serum creatinine < 1.5 mg/dL; WBC count >3,000/mm3, platelet count > 80,000/mm3, hemoglobin > 8 g/dL; total bilirubin value < 1.5 times the upper limit of normal [ULN], ALT level < 2.5 times ULN, AST < 2.5 times ULN.

Exclusion Criteria:

* pregnant or breast feeding
* a history of brain metastases or a primary brain tumor
* a history of hemorrhagic diathesis
* a history of corticosteroids or immunosuppressives use within four weeks of study entry
* a history of immune deficiency disorder or organ transplant
* has evidence of active adenovirus infection or uncontrolled infection
* received any chemotherapy or radiotherapy within four weeks of study entry

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2008-03; Primary Completion 2010-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
tumor response confirmed by CT or MRI | 3 months

SECONDARY OUTCOMES:
NCI toxicity criteria (CIC 3.0) | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Wenqi Jiang, Principal Investigator — Sun Yat-sen University
Locations (1):
- Cancer center, Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Lin X, Huang H, Li S, Li H, Li Y, Cao Y, Zhang D, Xia Y, Guo Y, Huang W, Jiang W. A phase I clinical trial of an adenovirus-mediated endostatin gene (E10A) in patients with solid tumors. Cancer Biol Ther. 2007 May;6(5):648-53. doi: 10.4161/cbt.6.5.4004. Epub 2007 Feb 13. PMID 17426445
- [Derived] Ye W, Liu R, Pan C, Jiang W, Zhang L, Guan Z, Wu J, Ying X, Li L, Li S, Tan W, Zeng M, Kang T, Liu Q, Thomas GR, Huang M, Deng W, Huang W. Multicenter randomized phase 2 clinical trial of a recombinant human endostatin adenovirus in patients with advanced head and neck carcinoma. Mol Ther. 2014 Jun;22(6):1221-1229. doi: 10.1038/mt.2014.53. Epub 2014 Mar 25. PMID 24662947